CLINICAL TRIAL: NCT03098914
Title: Clinical Characteristics and Microbiology of Community-Acquired Pneumonia: A Prospective Study
Brief Title: Clinical Characteristics and Microbiology of Community-Acquired Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Haidian Hospital (Other)
Collaborators: Beijing Tsinghua Chang Gung Hospital (Other); Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Liu chao, Doctor, Beijing Haidian Hospital
Other Study IDs: Beijing Haidian Hospital
Record Dates: First submitted 2017-03-22; First posted 2017-04-04 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Community-acquired Pneumonia
Keywords: Pathogen; Mortality; Community-acquired Pneumonia; Risk factors
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Beijing Haidian Hospital
  Interventions: Other: Cohort Study； pathogen； clinical features
- Chinese PLA General Hospital
  Interventions: Other: Cohort Study； pathogen； clinical features
- Beijing Tsinghua Chang gung Hospital
  Interventions: Other: Cohort Study； pathogen； clinical features

INTERVENTIONS:
Other: Cohort Study； pathogen； clinical features — Cohort Study； pathogen； clinical features

SUMMARY:
Community-Acquired Pneumonia has become common. Additionally, the mortality is high. But the epidemiology of pathogen is various in different areas, which is crucial for the key treatment. In addition, the risk factors of patients who died in 3 or 7 days in china is not clear, comparing with patients who died in 14 or 28 days or who survived.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed community acquired pneumonia
* Age≥18 ys

Exclusion Criteria:

* HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with commnuity acquired pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-04-11 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
the epidemiology of pathogen of community-acquired pneumonia in the three hospitals | confirmed as community-acquired pneumonia （2 weeks）
  screen out the pathogen of community-acquired pneumonia

SECONDARY OUTCOMES:
risk factors of patients who died in 3 or 7 days | in one week（3 days or 7days）
  patients who die in 3 or 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Haidian Hospital, Beijing, Beijing Municipality, China